CLINICAL TRIAL: NCT04315077
Title: The Effects of Short Term Oceanix Supplementation on Muscle Mass, Strength, and Power Underneath Extreme Training Conditions in Healthy and Elite Athletic Populations
Brief Title: The Short Term Effects of Oceanix Supplementation on Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Collaborators: Lonza Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0519
Record Dates: First submitted 2020-03-11; First posted 2020-03-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Oxidative Stress; Muscle Strength; Resistance Training; Muscle Damage; Immune Suppression
Keywords: Oxidative Stress; Muscle Strength; Antioxidants; Resistance Training; Immune Function; Exercise Recovery
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Double-Blind, Parallel, Randomized, Placebo-Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Subjects will consume one serving per day (25mg) of the treatment condition (Oceanix ®) for 21 days following baseline testing. Days 1 through 14 subjects will consume the supplement with the first meal of the day and refrain from resistance training. Days 15 through 19, subjects will complete one supervised resistance training each day and consume the supplement approximately 30 minutes prior to the training session. On days 20 and 21, subjects will complete follow-up testing in a manner identical to baseline and consume the supplement approximately 30 minutes prior to their arrival at the laboratory.
  Interventions: Dietary Supplement: Oceanix®; Other: Resistance Training
- Placebo Group (Placebo Comparator): Subjects will consume one serving per day (25mg) of the microcrystalline cellulose-based placebo condition for 21 days following baseline testing. Days 1 through 14 subjects will consume the supplement with the first meal of the day and refrain from resistance training. Days 15 through 19, subjects will complete one supervised resistance training each day and consume the supplement approximately 30 minutes prior to the training session. On days 20 and 21, subjects will complete follow-up testing in a manner identical to baseline and consume the supplement approximately 30 minutes prior to their arrival at the laboratory.
  Interventions: Other: Resistance Training

INTERVENTIONS:
Dietary Supplement: Oceanix® — Ingredient contains highly active antioxidant enzymes, including superoxide dismutase (SOD), as well as essential fatty acids, vitamins, amino acids and minerals.
  Arms: Experimental Group
Other: Resistance Training — 5 days of supervised and programmed whole-body resistance training.

SUMMARY:
The purpose of this study will be to examine the effects of Oceanix supplementation on isometric mid-thigh pull force kinetics and salivary immunoglobulin A (indice of immune function) following a one-week intense resistance training protocol. The study will be carried out in a randomized, double-blind, placebo-controlled, parallel manner. Subjects will be stratified into quartiles based on peak force achieved in the isometric mid-thigh pull assessment during screen and prior to baseline testing. Subjects from each quartile will be randomly divided by into treatment and or placebo conditions.

Following randomization, subjects will be baseline tested on isometric mid-thigh pull and salivary immunoglobulin A. Following baseline testing, subject will be given their respective supplement conditions and will be instructed to consume one serving (25mg) a day for 21 consecutive days. For days 1 through 14 subjects will be asked to refrain from resistance training. Subjects will undergo a five day intense resistance training protocol will on day 15 to day 19. Subjects will complete follow-up testing in a manner identical to baseline on day 20 and 21 (24- and 48-hours post completion of the training protocol).

DETAILED DESCRIPTION:
The purpose of this study will be to examine the effects of Oceanix supplementation on isometric mid-thigh pull force kinetics and salivary immunoglobulin A (indice of immune function) following a one-week intense resistance training protocol. The study will be carried out in a randomized, double-blind, placebo-controlled, parallel manner. Subjects will be stratified into quartiles based on peak force achieved in the isometric mid-thigh pull assessment during screen and prior to baseline testing. Subjects from each quartile will be randomly divided by into treatment and or placebo conditions. Supplement conditions will be provided in visually identical capsules and containers. Supplement compliance will be determined via supplement logs and collection of supplement containers on day 21. Subjects will be instructed to refrain from consuming other nutritional supplements for the duration of the study.

Following randomization, subjects will be baseline tested on isometric mid-thigh pull and salivary immunoglobulin A. Following baseline testing, subject will be given their respective supplement conditions and will be instructed to consume one serving (25mg) a day for 21 consecutive days. For days 1 through 14 subjects will be instructed to consume their condition with their first meal of the day, and they will asked to refrain from resistance training during this time frame. Subjects will undergo a five day intense resistance training protocol will on day 15 to day 19, and they will be instructed to consume their condition approximately 30 minutes prior to the training session. Subjects will complete follow-up testing in a manner identical to baseline on day 20 and 21 (24- and 48-hours post completion of the training protocol) consuming their condition approximately 30 minutes prior to their arrival at the laboratory.

The five day resistance training protocol will consist of two lower-, two upper-, and one full-body workout. Exercise sets performed on the first four days of the protocol will be targeted will repetition maximum loads such that sets will be perform to or near muscular failure. On the fifth day of the protocol, subjects will perform sets of bodyweight rear foot elevated split squats to failure for a total of 10 sets (5 sets with each leg in an alternating fashion). Subjects will be instructed to maintain the cadence set on an audible metronome, which will be set at one second downward and one second upward. Failure for these sets will be defined as 1) volitional muscle failure or 2) failure to complete two consecutive repetitions at the prescribed metronome cadence. Subjects will rest for one minute between sets. Prior to all training sessions, subjects will perform a dynamic warm-up, and following all training sessions, subjects will complete a cool down with static stretching of the targeted muscle groups with the session. All warm-up, resistance training, and cool down sessions will be supervised by trained research personnel. All training sessions will be separated by at least 24-hours.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 year of consistent resistance training experience (i.e. three days per week).
* Physically active males and females aged 18 to 45 years old.

Exclusion Criteria:

* Having a BMI of 30 or more kg/m²
* Having cardiovascular, metabolic, or endocrine disease.
* Undergone surgery that affects digestion and absorption.
* Smoker or use of smokeless tobacco
* Drinking heavily (> 7 and > 14 drinks per week for women and men, respectively).
* Women who are pregnant or planning to be pregnant.
* Taking medication to control blood pressure, lipids, and blood glucose
* Have taken or currently taking anabolic-androgenic steroids.
* Fish, shellfish, algae, or seaweed allergy.
* Any history of anabolic-androgenic steroid use.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Changes in Muscle Strength (Forces exerted in kg) | Baseline, 24-Hours Post Last Training Day, 48-Hours Post Last Training Day
  Assessed by Isometric Mid-Thigh Pull.
Changes in Rate of Force Development (Newtons per second) | Baseline, 24-Hours Post Last Training Day, 48-Hours Post Last Training Day
  Assessed by Isometric Mid-Thigh Pull

SECONDARY OUTCOMES:
Immunoglobulin A (micrograms per milliliter) | Baseline, 24-Hours Post Last Training Day, 48-Hours Post Last Training Day
  Experimental outcome examining the concentration of immunoglobulin A in fasted saliva sample.

OTHER OUTCOMES:
Repetitions Executed on a Bodyweight Rear Foot Elevated Split Squats | Fifth (Last) Day of Training Regimen.
  Recorded the number of repetitions executed.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Science & Performance Institute, Tampa, Florida, United States